CLINICAL TRIAL: NCT05947188
Title: A Prospective Multicenter Cohort Study for Non-invasive Diagnosis of Prostate Cancer: In Vivo Isolation of Circulating Tumor Cells Plus Multimodal MRI
Brief Title: Circulating Tumor Cells and mpMRI for Non-invasive Diagnosis of Prostate Cancer(CMNDPC)
Acronym: CMNDPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tianjin Medical University Second Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Affiliated Hospital of Nantong University (Other); Wujin People's Hospital (Other); Seventh Medical Center of PLA Army General Hospital (Other); The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XJTU1AF2022LSL-010
Record Dates: First submitted 2023-06-27; First posted 2023-07-17 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: Circulating Tumor Cells; multimodal MRI; Prostate Cancer; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample for Circulating Tumoral Cells (Experimental): Sampling of Circulating Tumoral Cells will be done
  Interventions: Other: prostate cancer diagnosis

INTERVENTIONS:
Other: prostate cancer diagnosis — prostate cancer diagnosis

SUMMARY:
This trial is a prospective, multicentre, diagnostic study. This study aims to evaluation the early diagnostic ability of circulating tumor cells plus multimodal MRI for prostate cancer.

DETAILED DESCRIPTION:
This trial is a prospective, multicentre, diagnostic study. This study aims to evaluation the early diagnostic ability of circulating tumor cells plus multimodal MRI for prostate cancer.

We will enroll 808 men with clinical suspicion of prostate cancer due to higher level PSA（>4ng/ml）or other examination abnormal. All the participants will receive prostate biopsy，the circulating tumor cells（CTCs）will be detected before biopsy.

This study will evaluate the diagnostic ability of CTCs+MRI and CTCs+MRI+PSA，including sensitivity, specificity, predictive values, diagnostic accuracy and receiver operating curves（ROC）.

ELIGIBILITY:
Inclusion Criteria:

1. No family history of prostate cancer;
2. men ≥ 50 years；
3. tPSA level of 4-10 ng/ml, and fPSA/tPSA<0.16;
4. tPSA level of >10 ng/ml；
5. With abnomal mpMRI、PET/CT、TRUS or DRE;
6. fully understand the clinical trial protocol and sign the informed consent;

Exclusion Criteria:

1. Not meet all of the inclusion criteria or any single inclusion criteria；
2. previous diagnosis of prostate carcinoma ;
3. symptomatic of acute prostatitis;
4. local anesthetic allergy patients;
5. cannot tolerate prostate biopsy or has contraindication to biopsy;
6. patients judged by the investigator to be unsuitable to participate in the clinical trial;

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of CTCs counts for prostate cancer | 12 weeks
  Evaluation the diagnostic ability of CTCs counts in caner and non-cancer. All patients were confirmed by pathology.

SECONDARY OUTCOMES:
Correlation between CTCs counts and PIRADS score | 12 weeks
  Diagnostic value of CTCs
combined PIRADS score for cancer and non-cancer | 12 weeks
  Diagnostic value of CTCs

CONTACTS AND LOCATIONS:
Overall Officials: yang gao, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: No